CLINICAL TRIAL: NCT04254822
Title: Hepatic Vein Pressure Gradient(HVPG)-Guided Therapy vs Carvedilol Plus Endotherapy for the Prevention of Esophageal Variceal Rebleeding in Patients With Liver Cirrhosis: A Prospective Randomized Controlled Trial
Brief Title: HVPG-Guided Therapy vs Carvedilol Plus Endotherapy for the Prevention of Esophageal Variceal Rebleeding in Cirrhotic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Tie Jun, Primary investigator, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY20192149-F-1
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Liver Cirrhoses; Variceal Hemorrhage; Esophageal Varices
Keywords: Transjugular intrahepatic portosystemic shunt; Endoscopic variceal ligation; Non-selective β-blocker therapy; Hepatic venous pressure gradient
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HVPG-guided therapy (Experimental): HVPG will be determined before randomization. In this arm, patients with an adequate reduction in HVPG (responders) receive carvedilol whereas nonresponders receive TIPS.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt; Drug: Carvedilol
- Standard therapy (Active Comparator): In this group, both responders and nonresponders will receive combination therapy of carvedilol and endoscopic variceal ligation as first-line therapy. If first-line therapy fails, TIPS will considered.
  Interventions: Drug: Carvedilol; Procedure: Endoscopic variceal ligation

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt — The TIPS procedures will be performed by experienced interventional radiologists. polytetrafluroethylene-covered stents were used with initial balloon dilatation to 8 mm, aiming for a decrease in portal-venous pressure gradient to less than 12 mm Hg.
  Arms: HVPG-guided therapy
Drug: Carvedilol — Carvedilol will be started at least 5 days after the index bleeding, unless a contraindication was present. Carvedilol will be start with 6.25 mg once a day and after 3 days increase to 6.25 mg twice-daily (the maximal dose was 12.5 mg/day). Systolic arterial blood pressure should not decrease <90 mmHg.
Procedure: Endoscopic variceal ligation — For endoscopic variceal ligation, the first elective session will be carried out within 7 days of randomisation. Then EBL sessions were scheduled every 10-14 days until variceal eradication (disappearance of varices or being too small to be sucked in the banding device).
  Arms: Standard therapy

SUMMARY:
Variceal bleeding is a major complication of cirrhosis, associated with a hospital mortality rate of 10%-20%. Surviving patients are at high risk for recurrent hemorrhage. For these reasons, management should be directed at its prevention. Endoscopic variceal band ligation (EBL) in combination with non-selective β-blocker (NSBB) therapy is the recommended first line therapy. Transjugular intrahepatic portosystemic stent-shunt (TIPS) is the most effective method to prevent rebleeding, however, it is burdened with increased hepatic encephalopathy and deterioration of liver function in patients with advanced cirrhosis. So TIPS placement forms an alternative if first line therapy fails.

Hepatic venous pressure gradient (HVPG) is currently the best available method to evaluate the presence and severity of portal hypertension. Patients who experience a reduction in HVPG of ≥20% or to <12mmHg in response to drug therapy are defined as 'responders'. The lowest rebleeding rates are observed in patients on secondary prophylaxis who are HVPG responders. A recent meta-analysis has demonstrated that combination therapy is only marginally more effective than drug therapy. This suggests that pharmacological therapy is the cornerstone of combination therapy. Adding EBL may not be the optimal approach to improve the outcome of HVPG nonresponders and HVPG non-responders are a special high-risk population that may benefit from a more aggressive approach, such as an early decision for TIPS. It recently was shown that TIPS placement within 72 hours after acute bleeding not only prevented recurrent bleeding but also improved survival. These raise the question of whether ligation together with NSBB should remain the first choice for elective secondary prophylaxis.

Therefore, the purpose of the study is to compare whether HVPG-guided therapy is superior to standard combination therapy for the prevention of variceal bleeding in patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of liver cirrhosis
* History of esophageal variceal bleeding confirmed by endoscopy
* Time interval between index bleeding and randomization > 5 days.
* Child-Pugh score < 12，MELD score<19

Exclusion Criteria:

* Clinical manifestation of active bleeding
* Gastric variceal bleeding: GOV2，IGV1 or IGV2
* Degree of main portal vein thrombosis > 50%
* Refractory ascites
* Contraindications of TIPS
* Contraindications of NSBB
* Budd-Chiari Syndrome
* Malignancy tumor
* Uncontrolled infections
* History of portal-systemic shunt surgery
* HIV
* Pregnancy or breastfeeding woman
* Poor incompliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of esophageal variceal rebleeding | 12 months
  Source of variceal rebleeding will be determined by endoscopy.

SECONDARY OUTCOMES:
Cumulative incidence of variceal rebleeding related death | 12 months
Cumulative incidence of all cause mortality | 12 months
Cumulative incidence of patients with further decompensation | 12 months
  Decompensation was defined as variceal rebleeding, ascites, and hepatic encephalopathy
Cumulative incidence of patients with ascites | 12 months
Cumulative incidence of patients with hepatic encephalopathy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jun Tie, M.D.,Ph.D., Principal Investigator — Air Force Military Medical University, China
Locations (1):
- Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No